CLINICAL TRIAL: NCT02144272
Title: A Phase 1 Single-Dose, Dose Escalation Study to Evaluate the Safety and Tolerability of LY3114062 in Subjects With Inflammatory Arthritis
Brief Title: Safety Study to Evaluate LY3114062 in Participants With Inflammatory Arthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 15098; I6W-MC-TNAA (Other: Eli Lilly and Company)
Record Dates: First submitted 2014-05-19; First posted 2014-05-21 (Estimated); Last update posted 2015-07-17 (Estimated); Status verified 2015-07

CONDITIONS: Inflammatory Arthritis
Keywords: Antibody; Tumor Necrosis Factor alpha; Interleukin-17
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- LY3114062 (SC) (Experimental): LY3114062 given as a single subcutaneous (SC) dose, in escalating dose cohorts starting at 2 mg.
  Interventions: Drug: LY3114062 SC
- LY3114062 (IV) (Experimental): LY3114062 given once intravenous (IV).
  Interventions: Drug: LY3114062 IV
- Placebo (Placebo Comparator): Placebo (sodium chloride injection) given as a single SC dose.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3114062 SC — LY3114062 administered SC.
  Arms: LY3114062 (SC)
Drug: Placebo — Placebo administered SC.
  Arms: Placebo
Drug: LY3114062 IV — LY3114062 administered IV.
  Arms: LY3114062 (IV)

SUMMARY:
The main purpose of this study is to learn more about the safety of LY3114062 and to find out how well it is tolerated in participants with an inflammatory arthritis. The study will also investigate how the body processes the drug and how the drug affects inflammatory arthritis. The study is expected to last about 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Signs or symptoms of an inflammatory arthritis for a duration of at least 8 weeks at screening.
* Presence of at least 3 out of 66 swollen joints at screening and baseline, as determined by the swollen joint count assessment forms.

Exclusion Criteria:

* Synthetic disease-modifying antirheumatic drugs DMARD use as follows:

  * ANY treatment with tofacitinib within 28 days prior to baseline or planned treatment with tofacitinib during the study;
  * Treatment with other synthetic DMARDs (eg, hydroxychloroquine, methothrexate, leflunomide, sulfasalazine, and gold salts) at an unstable dose within 28 days prior to baseline or if the dose of drug is planned to be changed during the study.
* Previous treatment with marketed biologic DMARDs as follows:

  * Etanercept, adalimumab, or anakinra <4 weeks prior to baseline;
  * Infliximab, certolizumab pegol, golimumab, abatacept, or tocilizumab <8 weeks prior to baseline;
  * Rituximab <12 months prior to baseline

Note: Other biologic agents for indications other than an inflammatory arthritis may be allowed after discussion with the sponsor

* Treatment with >10 mg/day, or unstable dose, of oral prednisone or equivalent within 28 days prior to baseline.
* Confirmed or suspected septic arthritis, crystal arthropathy, systemic lupus erythematosus, reactive arthritis, or certain other rheumatic conditions.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2014-06; Primary Completion 2015-05 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
The Number of Participants with One or More Drug-Related Adverse Events | Baseline to study completion (3 months)

SECONDARY OUTCOMES:
Pharmacokinetics: Maximum Plasma Concentration (Cmax) of LY3114062 | Predose through Day 85, at specified timepoints
Pharmacokinetics: Area Under the Concentration-time curve (AUC) of LY3114062 | Predose through Day 85, at specified timepoints
Antibody Production Against LY3114062 | Day 1, 8, 15, 29, 85 and early discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9 AM-5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (4):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sofia, Bulgaria
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tbilisi, Georgia
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chisinau, Moldova
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bucharest, Romania